CLINICAL TRIAL: NCT03104829
Title: A Randomized Control Trial Compare Between Diabetic Knowledge and Self-care Behaviors (DSME) With and Without Motivational Interviewing, on Glycemic Control Among Children and Adolescents With Diabetes Mellitus Type 1
Brief Title: DSME or DSME + MI in T1DM on Glycemic Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-DSME-MI-01
Record Dates: First submitted 2017-03-26; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DSME (Active Comparator): participants in this arm will receive standard care for diabetes (DSME) at the beginning of the study and 3 months later
  Interventions: Drug: DSME participants in this arm will receive standard care for diabetes (DSME) at the beginning of the study and 3 months later
- DSME+MI (Experimental): participants in this arm will receive standard care for diabetes plus motivation interviewing (MI) sessions at the beginning of the study and 3 months later, will also receive motivation interviewing sessions by phone at 1, 2, 4, 5 month after the beginning of the study
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing
  Arms: DSME+MI
Drug: DSME participants in this arm will receive standard care for diabetes (DSME) at the beginning of the study and 3 months later
  Arms: DSME

SUMMARY:
This study evaluates the effect of diabetic knowledge and self care behavior (DSME) alone or DSME plus motivational interviewing on glycemic control among children and adolescents with DM type 1. Half of participants will receive DSME along, while the other half will receive DSME plus MI.

ELIGIBILITY:
Inclusion Criteria:

* T1DM
* age more than 10 years old
* HbA1C more than 8%

Exclusion Criteria:

* other types of DM
* receive medications that may effect blood glucose
* mental retardation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
HbA1C | at the beginning of the study, 3 month and 6 months later

SECONDARY OUTCOMES:
Pre and post test scores for Diabetic knowledge | at the beginning and 6 months later
Diabetic self-care behavior score | at the beginning and 6 months later

CONTACTS AND LOCATIONS:
Overall Officials: Ornsuda Lertbannaphong, MD, Principal Investigator — Endocrinology Division, Pediatrics department, Siriraj Hospital
Locations (1):
- Ornsuda Lertbannaphong, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Santiprabhob J, Likitmaskul S, Kiattisakthavee P, Weerakulwattana P, Chaichanwattanakul K, Nakavachara P, Peerapatdit T, Nitiyanant W. Glycemic control and the psychosocial benefits gained by patients with type 1 diabetes mellitus attending the diabetes camp. Patient Educ Couns. 2008 Oct;73(1):60-6. doi: 10.1016/j.pec.2008.05.023. Epub 2008 Jul 7. PMID 18606522
- [Background] Viner RM, Christie D, Taylor V, Hey S. Motivational/solution-focused intervention improves HbA1c in adolescents with Type 1 diabetes: a pilot study. Diabet Med. 2003 Sep;20(9):739-42. doi: 10.1046/j.1464-5491.2003.00995.x. PMID 12925054